CLINICAL TRIAL: NCT06649097
Title: Clearance of Intracranial Blood Products by Continuous Irrigation With the IRRAflow System
Acronym: CRYSTAL
Status: Recruiting | Type: Observational
Sponsor: Christopher P Kellner (Other)
Collaborators: IRRAS (Industry)
Responsible Party: Sponsor-Investigator, Christopher P Kellner, Associate Professor, Neurosurgery, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Other Study IDs: STUDY-24-01230
Record Dates: First submitted 2024-10-16; First posted 2024-10-18 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Intracranial Hemorrhage; Ventriculitis; Intracranial Abscess
MeSH Terms: conditions — Intracranial Hemorrhages | interventions — Drug Delivery Systems

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- IRRAflow device: All patients enrolled into the study will undergo treatment with the IRRAflow device
  Interventions: Device: IRRAflow® CNS (Active Fluid Exchange) System

INTERVENTIONS:
Device: IRRAflow® CNS (Active Fluid Exchange) System — The IRRAflow system offers automated irrigation, controlled drainage and intracranial pressure (ICP) monitoring all in one system. It consists of three main parts - IRRAflow 2.0 Catheter, IRRAflow Tube Set, IRRAflow Control Unit.

SUMMARY:
The study is a multi-center prospective cohort, controlled, phase 4 post-market registry evaluating the efficacy and radiographic outcomes associated with the use of the IRRAflow® Active Fluid Exchange System compared to standard of care external ventricular drains.

DETAILED DESCRIPTION:
The IRRAflow system offers automated irrigation, controlled drainage, and ICP monitoring all in one system for the treatment of intracranial hemorrhage - [Intracerebral hemorrhage (ICH), Intraventricular hemorrhage (IVH), Subarachnoid hemorrhage (SAH), Subdural hematoma (SDH)], intracranial abscess, and ventriculitis.

The analysis of the IRRAS catheter will occur prospectively if it is determined the patient meets the enrollment criteria. All patients enrolled in the trial will receive additional supportive and medical treatment by choice of the treating physician and in accordance with standard of care. Such treatment includes but is not limited to neurointensive care, neuromonitoring, and surgical or endovascular occlusion of identified sources of intracranial hemorrhage (e.g. vascular anomalies, aneurysms, etc.).

ELIGIBILITY:
Inclusion criteria:

* Age >=18 years of age
* Intracranial hemorrhage documented on head CT or MRI scan.
* Indication for active fluid exchange evaluated by treating physician.
* Signed informed consent obtained by patient or Legal Authorized Representative
* Scheduled enrollment and treatment within 72 hours of last known well (LKW)

Exclusion criteria:

* GCS ≤ 5
* Pregnancy
* Fixed and dilated pupil
* Life-threatening medical condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient population for this study will be comprised of up to 250 patients with primary diagnosis of intracranial hemorrhage (SAH, ICH, IVH, SDH), ventriculitis, or intracranial abscess.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-09-25 (Actual); Primary Completion 2031-01 (Estimated); Study Completion 2031-07 (Estimated)

PRIMARY OUTCOMES:
Residual blood volume by post bleed day 5 | Post-procedure day 5
  The residual blood volume at day 5 will be calculated to determine the efficacy of the IRRAflow system compared to other external ventricular drains (EVDs)
Utility weighted modified Rankin Score | End of study, at 6 months
  Modified Rankin Scale score at 6 months will be collected to determine patient functional outcomes at 6 months. Scores range from 0 to 6, with 0 indicating no disability and 6 indicating death

SECONDARY OUTCOMES:
Rate of blood clearance | Immediately before and after the procedure
  Rate of blood clearance will be calculated based on pre- and post-procedure blood volumes
Direct hospitalization costs | Discharge, up to 7 days post procedure
  Direct hospitalization costs will be determined based on the hospital-reported cost of care for the entirety of the patient's hospital stay
NSICU Length of Stay | Discharge, up to 7 days post procedure
  Hospital quality metrics will include length of neonatal surgery intensive care unit (NSICU) stay in days
Hospital Length of Stay (LOS) | Discharge, up to 7 days post procedure
  Hospital quality metrics will include length of hospital stay in days
Proportion of participants needing a shunt | Discharge, up to 7 days post procedure
  Proportion of participants needing a shunt will be calculated to determine how many patients needed a shunt to treat their hydrocephalus

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Kellner, Principal Investigator — Icahn School of Medicine at Mount Sinai; Nicholas Brandmeir, Principal Investigator — West Virginia University
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Upon the completion of the study, Mount Sinai's data management team will clean and analyze all data in preparation of manuscript writing and publication. The intention will be to publish together between the principal investigator and the sponsor. Following publication, Mount Sinai will archive and store all associated data on its cloud-based system.